CLINICAL TRIAL: NCT06247176
Title: Neurobiological Mechanisms of Sensory Hyper-sensitivity and Habituation in Autism Spectrum Disorders
Brief Title: Sensory Habituation in Autism Spectrum Disorders
Acronym: ASD_VR_RE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI no longer at institution.
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 0709-22-EP
Record Dates: First submitted 2024-01-22; First posted 2024-02-07 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Autism Spectrum Disorder; Autism; Sensory Processing Disorder; Sensory Over-Responsivity
Keywords: Autism; Autism Spectrum Disorder; Virtual Reality; Sensory Sensitivity; Sensory Hyper-reactivity; Sensory Processing; Sensory Over-Responsivity
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder

STUDY DESIGN:
Intervention Model Description: There will be two groups, one group will be subjects with autism spectrum disorder and the second group will be subjects who are neurotypical. Each group will participate in the same habituation protocol.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Autism Spectrum Disorder Habituation Group (Experimental): This will be the group of subjects with Autism and sensory over-responsivity. This group will go through a mock-MRI, a pre-habituation MRI, the habituation protocol in virtual reality, and a post-habituation MRI.
  Interventions: Behavioral: Sensory Habituation Protocol
- Neurotypical Habitation Group (Active Comparator): This will be the group of subjects who are neurotypical peers. This group will go through a mock-MRI, a pre-habituation MRI, the habituation protocol in virtual reality, and a post-habituation MRI.
  Interventions: Behavioral: Sensory Habituation Protocol

INTERVENTIONS:
Behavioral: Sensory Habituation Protocol — The first session continues with the Mock MRI, which lasts 10 minutes. Participant's comfort level in VR will be evaluated.
  At the pre-exposure visit, participants complete an MRI scan on a 3 Tesla MRI, which takes approximately 1 hour & 15 minutes. It consists of structural & functional MRI scans. Structural scans require the participant to stay still with eyes closed. Functional scans will require the participant to lie with eyes closed or watch and listen to sensory stimulation.
  VR exposure will occur across 3 1-hour sessions at most. Participants will be asked to complete a sensory habituation protocol, in which they will watch and listen to sensory stimuli in VR for an increasing amount of time. Between the sensory stimuli, the participant will watch a self-selected video.
  Finally, the subject will be asked to do a post-exposure MRI visit, which is the same as the pre-exposure visit.
  Other Names: Repeated Exposure

SUMMARY:
Autism spectrum disorder (ASD) is one of the most common developmental disabilities and often people with ASD have sensory processing disorders. These sensory processing disorders are often associated with problem behaviors and, more recently, have been connected to anxiety disorders in people with ASD. While it has been suggested that sensory processing responses in ASD could be malleable, current treatment strategies for sensory processing disorders in ASD have inconsistent results or lack large-sample sized data. This investigation will explore changes in neurophysiological activity in people with ASD and neurotypical peers after they are exposed to an unpleasant visual stimulus through a virtual reality systematic desensitization protocol. 30 people with ASD and 30 neurotypical people between the ages 7 - 35 will be recruited. The study have, 1) a practice magnetic resonance imaging (MRI) visit with questionnaires, 2) a per-exposure MRI with structural and functional MRI collections, 3) a virtual reality systematic desensitization session where we will record the participant's physiological response using an Emotibit device, and 4) a post-exposure MRI session with structural and functional MRI collections. This investigation aims to quantify changes in neurophysiological responses in order to determine the effect of systematic desensitization.

DETAILED DESCRIPTION:
Autism Spectrum Disorder (ASD) is one of the most common developmental disabilities, with an estimated 1 in 54 children receiving a diagnosis. The total economic burden of ASD in the United States is estimated to be $268 billion and will increase to $461 billion by 2025. People with ASD have deficiencies in social relationships and communications and an increased rate of anxiety disorders, with some estimates suggesting 84% of people with ASD have anxiety. This anxiety can lead to an individual with ASD to exhibit avoidant behavior, which can include exclusion from activities to escalated behaviors that could be self-injurious or harmful to others. These avoidant behaviors can make participation in activities of daily living challenging for people with ASD, as the avoidant behavior is often considered socially-unacceptable behavior. While there has been increasing interest in anxiety in ASD, there is still a major knowledge gap in understanding how sensory processing disorders play a role in anxiety and if this can be treated.

Sensory Processing in ASD: Sensory processing disorders were added to ASD diagnosis in The Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition in 2013. Since then, there has been little research into the role that sensory processing disorders plays in the anxiety of people with ASD. Functional magnetic resonance imaging (fMRI) studies have demonstrated that people with ASD have greater brain activity in relevant sensory areas, the amygdala, and the orbital frontal cortex when exposed to combinations of unpleasant auditory, tactile, or visual stimuli. Further, people with ASD have a reduced ability to habituate to the same unpleasant stimuli in the relevant sensory cortices and amygdala, differences in the changes of brain activity in the orbital-frontal cortex, and differences in functional connectivity between the amygdala and orbital-frontal cortex. These brain responses have also been connected with physiological responses in children with ASD, as those with greater skin conductivity having reduced neural response in the orbital-frontal cortex and heart rate being positively correlated with activity in the inferior and medial frontal gyrus.

Even though the neurophysiological evidence supports sensory processing differences in ASD, current treatment strategies are sparse and the results are often inconsistent. The most successful paradigm is exposure therapy through systematic desensitization, which has been used in both ASD and people with anxiety. While multisensory integration skills may be malleable, it has been suggested that exposure therapy may not be an effective long-term strategy, as the clinical team cannot perform exposure to every stimulus in every environment. With this in mind, new therapeutic techniques need to be designed to enable personalization of exposure experiences.

Virtual Reality for ASD: One emerging technique that could enable quick personalization of unpleasant stimulus and environments is virtual reality (VR). Therapeutic VR software has shown to be an effective platform for skill training, mainly focusing on behavioral skills in social or educational environments. Two investigations demonstrated changes in neural activity after participating in VR social cognition training. However, the effects of using VR as a sensory exposure platform on the physiological response to unpleasant stimuli has not been explored.

Purpose The research objectives of this application are to quantify the neurophysiological changes that occur after participating in a virtual reality systematic desensitization protocol. The following aims will be achieved the top physiological recording devices for ASD to collect physiological responses, front-line virtual reality systems to provide automated desensitization exposure therapy, and University of Nebraska Medical Center's research MRI system. 30 people with ASD and 30 neurotypical peers will be recruited to utilize this software. This proposal will be the first step in developing evidence-based therapies aimed at addressing sensory processing differences in ASD.

ELIGIBILITY:
Inclusion Criteria:

* For our patient population

  1. people with a diagnosis of autism spectrum disorder
  2. people who have sensory over-responsivity
  3. can wear a VR headset for up to 20 minutes
  4. can understand and follow directions

For neurotypical participants

1. can wear a VR headset for up to 20 minutes
2. can understand and follow directions

Exclusion Criteria:

* 1) if you have any known visual impairment that will make it difficult to watch an object in a VR headset 2) inability to wear a VR headset 3) a history of seizures 4) A subject with orthodontic braces or metallic implants, such as prostheses, shrapnel, or aneurysm clips, or persons with electronic implants, such as cardiac pacemakers. The magnetic field generated by the MRI machine can cause a displacement or malfunctioning of these devices; 5) A subject who is claustrophobic, unable to stay still in the scanner for 40 minutes, or unable to be in the MRI scanner room alone;

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1 (Actual)
Dates: Start 2024-01-08 (Actual); Primary Completion 2024-10-07 (Actual); Study Completion 2024-10-07 (Actual)

PRIMARY OUTCOMES:
Changes in neural response to the sensory stimulation | There are two 1 hour sessions in which the bold response will be measured. The first time point will be during visit 2 of the study. The second time point will be the final visit of the study.
  This will be the change in the bold response as measured by the fMRI scan.

SECONDARY OUTCOMES:
Galvanic Skin Response as measured by a physiological recording devices, either an Emotibit or the MRI scanner | Galvanic skin response will be measured at 3 - 5 time points, ranging from 1 hour and 30 minutes to 3 hours and 30 minutes of data. 15 minutes will be measured at the 2nd and last visit. 1 hour will be collected at each VR visit.
  Galvanic skin response is a measure of how sweaty the skin is and can be used as a measure of the body's stress. We will look at this before during and after the habituation protocol to measure how the body adapts to the sensory stimulation.
Changes in skin temperature after going through a sensory habituation protocol, measured by an Emotibit | Skin temperature will be measured at 1 - 3 time points, ranging from 1 hour to 3 hours of data. 1 hour will be collected at each VR visit.
  This will look at the change in the skins temperature before, during, and after the sensory habituation protocol. This is a measure of the body's response to a stressor.
Heart rate changes as measured by a physiological recording devices, either an Emotibit or the MRI scanner | Heart rate will be measured at 3 - 5 time points, ranging from 1 hour and 30 minutes to 3 hours and 30 minutes of data. 15 minutes will be measured at the 2nd and last visit. 1 hour will be collected at each VR visit.
  Changes in heart rate can give an indication of stress and habituation. This will be recorded before, during, and after the habituation protocol to assess how the body reacts.

CONTACTS AND LOCATIONS:
Overall Officials: James E Gehringer, PhD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Munroe-Meyer Insitute, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified MRI scans and physiological responses will be made available after completion of the study.
Supporting Information: Study Protocol
Time Frame: De-identified data will be released after conclusion of data collections (planned for end of 2025), conclusion of data analysis (planned for end of 2026), and submission of publication (planned for end of 2026/early 2027)
Access Criteria: Data will be made available upon reasonable request.
URL: https://www.unmc.edu/mmi/research/virtual-reality-lab.html